CLINICAL TRIAL: NCT01542944
Title: TevaGastrim for Stem Cell Mobilization of HLA Matched Sibling Donors for Allogeneic Hematopoietic Stem Cell Transplantation in Patients With Acute Myelogenous Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Brief Title: TevaGastrim for Stem Cell Mobilization Sibling Donors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-11-9090-AN-CTIL
Record Dates: First submitted 2012-02-19; First posted 2012-03-02 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Acute myeloid leukemia; Myelodysplastic syndrome; Stem Cell Mobilization; Allogeneic Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TevaGastrim (Experimental): treatment with TevaGastrim for allogeneic stem cell collection
  Interventions: Drug: TevaGastrim

INTERVENTIONS:
Drug: TevaGastrim — TevaGastrim 10 mg/kg SC will be administered in the evening for 4 days prior to apheresis.

SUMMARY:
The aim of this study is to evaluate the efficacy of TevaGastrim which is a biosimilar version of Filgrastim recombinant human G-CSF (G-CSF) in mobilizing sufficient number of stem cells from normal sibling donors for allogeneic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years.
2. Normal sibling donor that is HLA matched to a patient with AML or MDS that needs and is eligible for allogeneic stem cell transplantation
3. Written informed consent.

Exclusion Criteria:

1. Inability to tolerate PBPC harvest.
2. Peripheral venous access not possible.
3. Positive pregnancy test for female donors.
4. Positive serology for hepatitis C and/or HBSAg, unless negative for antigen PCR.
5. Psychiatric, addictive, or any disorder which compromises ability to give truly informed consent for participation in this study.
6. Treatment with other investigational drugs.
7. Known sensitivity to CHO derived products.
8. HIV positive.
9. History of malignant disease or current malignancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Mobilisation success rate | 4 weeks
  Mobilisation success rate is defined as the mobilisation of a PBSC graft containing >2x106 CD34+ cells/kg in ≤ 4 apheresis sessions. We will evaluate the time from chemotherapy to stem cell collection,number of collections required to reach >2x106 CD34+ cells/kg, number of CD34+ cells collected and percentage of patients reaching >5x10 CD34+ cells/kg in ≤ 4 apheresis sessions.

SECONDARY OUTCOMES:
engraftment after transplantation | 100 days
  speed of engraftment is determined by the time until recovery of blood counts after transplantation
Donor safety | 100 days
  To determine side effects to the stem cell donor

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel